CLINICAL TRIAL: NCT00945958
Title: Evaluation of Safety of SPARC0913 in Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLR_09_13
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2016-05

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPARC0913 (Experimental)
  Interventions: Drug: SPARC0913

INTERVENTIONS:
Drug: SPARC0913 — One drop of SPARC0913 in affected eye once daily for 24 weeks

SUMMARY:
The purpose of this study is to evaluate the long-term safety of SPARC0913. A multicenter, open label, non-randomized, uncontrolled, single group assignment, safety study of subjects with primary open angle glaucoma or ocular hypertension is planned. Subjects will receive study medication for a period of 24-weeks.

DETAILED DESCRIPTION:
This is a multicenter, open label, non-randomized, single-arm, extension safety study to evaluate the long-term safety of SPARC0913. Subjects who completed the prior evaluator-masked clinical non-inferiority Study participated in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years
* Willing to participate and giving written informed consent
* Willing to commit to study medication-dosing, study visits and follow-up visits to complete evaluation
* Eligible to receive Latanoprost once a daily as monotherapy for treatment of glaucoma

Exclusion Criteria:

* History of allergic hypersensitivity or poor tolerance to latanoprost
* History of Substance abuse or addiction (alcohol drugs) in the past 3 years
* History of chronic use of concomitant medications in neurologic or psychiatric illness that would affect assessment of safety and effectiveness of the study medication
* Any abnormality preventing IOP measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC study site, High Point, North Carolina, United States

REFERENCES:
- [Derived] Shen Lee B, Malhotra R, Sall K, Mitchell B, Peace J. Open-Label Extension Study Comparing Latanoprost 0.005% Without vs With Benzalkonium Chloride in Open-Angle Glaucoma or Ocular Hypertension. Clin Ophthalmol. 2022 Jul 19;16:2285-2293. doi: 10.2147/OPTH.S367756. eCollection 2022. PMID 35898518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an extension study of previous study conducted by SPARC (CLR_09_12).
  This was open-label, single group assignment long-term safety study.
  A total of 161 subjects were enrolled in this study.
  From the start of the study through Week 24 (Visit 7), safety endpoints (TEAEs and change introocular pressure) were evaluated
Pre-assignment Details: Subjects received their first dose of the study drug at Visit 1 (Baseline Visit). A total of 149 subjects completed Study Visit 7 (End-of-Evaluations), which met FDA's recommendation of providing safety data for at least 100 subjects for at least 6 months.
Period: Overall Study
Arm/Group | SPARC0913
Started | 161
Completed | 149
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: A total of 161 subjects enrolled in the study. Subjects received their first dose of the study drug at Visit 1 (Baseline Visit). A total of 149 subjects completed Study Visit 7 (End-of-Evaluations), which met FDA's recommendation of providing safety data for at least 100 subjects.
Groups:
- SPARC0913: Inhaled dose of SPARC0913. Each single dose was administered as 1, 2, 4 and 8 puffs from the inhaler.
Arm/Group | SPARC0913
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With AEs
Description: Subjects with treatment emergent adverse events
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- SPARC: The number and percentage of subjects reporting a TEAE were tabulated by system organ classification and preferred terms.
Arm/Group | SPARC
Number analyzed (Participants) | 161
participants | 140

2. Secondary Outcome: Mean Change in IOP From Baseline to Visit 7 (End of Evaluations Visit)
Description: From the start of study (baseline visit) through week 24 (Visit 7, end of evaluations visit), the change in IOP was measured
Time Frame: 24 weeks
Population: From the start of the study through Week 24 (Visit 7, End of Evaluations), the change in IOP is evaluated
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | SPARC0913
Number analyzed (Participants) | 161
mm Hg | 2.83 (4.20)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Of the 161 enrolled subjects in the study, 149 subjects received at least 24 weeks of SPARC's latanoprost treatment (completed the End-of-Evaluations i.e. Week 24), which met FDA's recommendation of providing safety data for at least 100 subjects.
Groups:
- SPARC0913: From the start of the study through Week 24 (Visit 7, End of Evaluations) adverse events were evaluated
Arm/Group | SPARC0913
Serious Adverse Events (participants affected / at risk) | 5/161
Other Adverse Events (participants affected / at risk) | 140/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPARC0913 (N=161)
Peripheral vascular disease (Vascular disorders) | 1 (1)
Acute tension headache (Nervous system disorders) | 1 (1)
Epididymitis orchitis (Infections and infestations) | 1 (1)
Carotid stenosis (Nervous system disorders) | 1 (1)
Syncopal episode (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPARC0913 (N=161)
Influenza, Sinusitis, Conjunctivitis viral, Tooth infection (Infections and infestations) | 12 (15)
Dizziness,Visual field defect (Nervous system disorders) | 6 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0)
Edema peripheral (General disorders) | 2 (2)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Any PT (Metabolism and nutrition disorders) | 2 (5)
any PT (Psychiatric disorders) | 1 (1)
Eye pain, ocular hyperemia, growh of eyelashes (Eye disorders) | 140 (319) — eyelash thickening, eye discharge, conjunctival hyperemia, erythema of eyelid, punctate keratitis, visual acuity reduced, dry eye, cataract, conjunctival hemorrhage, eyelash discoloration, vitreous detachment, conjunctival edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other